CLINICAL TRIAL: NCT02551003
Title: A Multi-Centre Safety and Efficacy Study of Autologous Cord Blood Combined With Therapeutic Hypothermia Following Neonates Encephalopathy in China
Brief Title: Neuroprotective Effect of Autologous Cord Blood Combined With Therapeutic Hypothermia Following Neonatal Encephalopathy
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study did not commence due to unforeseen challenges in securing adequate funding and resources, coupled with logistical constraints.
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Maternal and Child Health Hospital of Guangxi Zhuang Autonomous Region (Other); Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHFudanU_NNICU1; NCT02605018 (obsolete NCT alias)
Record Dates: First submitted 2015-09-04; First posted 2015-09-16 (Estimated); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Hypoxic Ischemic Encephalopathy; Cerebral Infarction
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Cerebral Infarction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cord blood with hypothermia (Experimental): Autologous cord blood will be collected after birth and stored in Cord Blood Bank of hospital. All cord blood samples are routinely performed by dedicated, trained UCB collection staff and is restricted to deliveries of mothers who have given prior written informed consent for collection. If the mother delivered a baby with signs of HIE or cerebral infarction, Bank staff collected UCB utilizing standard procedures. Collected UCB was transported at roomtemperature in validated shippers to the NICU. Infusions were started when cells and study staff were available for administration and monitoring. Infants received up to 3 infusions, with the first dose as soon as possible after birth, and at, 48, and 72 postnatal hours. At the same time, babies will referred to neonatal intensive care unit for hypothermia therapy of cooling to 33.5 ℃ body temperature for 72 hours and standard intensive care.
  Interventions: Drug: Autologous cord blood
- Hypothermia (Active Comparator): Hypothermia therapy of cooling to 33.5 ℃ body temperature for 72 hours and standard intensive care.
  Interventions: Device: Hypothermia

INTERVENTIONS:
Drug: Autologous cord blood — Autologous cord blood will be collected after birth and administered in divided aliquots during the first 3 days of life. At the same time, babies will referred to neonatal intensive care unit for hypothermia therapy of cooling to 33.5 ℃ body temperature for 72 hours and standard intensive care.
  Arms: Cord blood with hypothermia
Device: Hypothermia — Hypothermia therapy of cooling to 33.5 ℃ body temperature for 72 hours and standard intensive care.
  Arms: Hypothermia

SUMMARY:
This study examines the effect of cord blood in the treatment of newborn infants with neonatal encephalopathy in combination with hypothermia, which is the standard treatment for this condition. The hypothesis is that the cord blood + hypothermia combination will produce better neuroprotection than the standard treatment of hypothermia alone.

DETAILED DESCRIPTION:
The primary aim of this study is to determine the neuroprotective effect of intravenous administration of autologous cord blood in neonates with severe encephalopathy (hypoxic ischemic encephalopathy or cerebral infarction). It is hypothesized that the administration of autologous cord blood will be safe and well tolerated in neonates with severe encephalopathy. If a neonate is born with signs of moderate to severe encephalopathy and cooled for the encephalopathy, the neonate will receive their own cord blood. The cord blood cells are divided into 3 doses and infused at 24, 48, and 72 hours after the birth. Infants will be randomised to treatment with autologous cord blood and hypothermia or hypothermia only and followed for safety and neurodevelopmental outcome up to 18 months. All infants in both groups will be treated with hypothermia for 72 hours started within 6 hours of delivery and infants who allocated to hypothermia and xenon will also receive autologous cord blood in 24 hours from birth through a purpose designed delivery system. Additionally, postnatal neuro-developmental outcomes in neonates with encephalopathy after autologous cord blood therapy will be measured; HIE injury to the neonate/infant brain post autologous cord blood therapy by imaging will be characterized; MRI's will be obtained per clinical routine; serum levels of selected cytokine and neurotrophic factors in neonates with HIE before and after autologous cord blood therapy will be compared and immune cell phenotype and function in neonates with HIE before and after autologous cord blood therapy will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age ≥ 34 weeks
2. Birth weight ≥ 1800 grams
3. 10-minute Apgar score ≤5 or continued need for ventilation or severe acidosis, defined as pH <7.0
4. Moderate to severe encephalopathy (Sarnat II to III)
5. A moderately or severely abnormal background aEEG voltage, or seizures identified by aEEG, if monitored
6. Up to 24 hours of age
7. Autologous umbilical cord blood available to infuse 3 doses within 72 hours after birth
8. Parental informed consent

Exclusion Criteria:

1. Known major congenital anomalies, such as chromosomal anomalies, heart diseases
2. Major intracranial hemorrhage identified by brain ultrasonography or computed tomography
3. Severe intrauterine growth restriction (weight <1800g)
4. Severe infectious disease, such as sepsis
5. Inability to enroll by 24 hours of age
6. Volume of collected cord blood <40 ml
7. Infants in extremis for whom no additional intensive therapy will be offered by attending neonatologist
8. Parents refuse consent

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2015-09-08 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Mortality | From birth to the age of 18 months
  The relative frequency of deaths in each group.
Disability Rate | From birth to the age of 18 months
  Disability, defined as a physical or mental handicap, especially one that prevents a person from living a full, normal life or from holding a gainful job.

SECONDARY OUTCOMES:
Neurodevelopment(Bayley Scores) | At the age of 12 months
  Efficacy of levetiracetam by assessment of the change from baseline to 12 months in neurodevelopment via Bayley Scores of Infant Development Mental Development Index (BSID).
Neurodevelopment(Bayley Scores) | At the age of 18 months
  Efficacy of levetiracetam by assessment of the change from baseline to 18 months in neurodevelopment via Bayley Scores of Infant Development Mental Development Index (BSID).
Brain Structural Alterations(MRI) | At the age of 7 days
  Efficacy of cord blood by assessment of the changes in brain from baseline in MRI on Day 7.
Brain Structural Alterations(MRI) | At the age of 28 days
  Efficacy of cord blood by assessment of the changes in brain from baseline in MRI on Day 28.
Brain Structural Alterations(MRI) | At the age of 12 months
  Efficacy of cord blood by assessment of the changes in brain from baseline in MRI on 12 months old.
Brain Parenchyma Alterations(MRI) | At the age of 7 Days
  Efficacy of cord blood by assessment of the changes in brain from baseline in MRI on Day 7.
Brain Parenchyma Alterations(MRI) | At the age of 28 days
  Efficacy of cord blood by assessment of the changes in brain from baseline in MRI on Day 28.
Brain Parenchyma Alterations(MRI) | At the age of 12 months
  Efficacy of cord blood by assessment of the changes in brain from baseline in MRI on 12 months old.
Intracranial Hemorrhage(MRI) | At the age of 7 days
  Efficacy of cord blood by assessment of the changes in brain from baseline in MRI on Day 7.
Intracranial Hemorrhage(MRI) | At the age of Day 28
  Efficacy of cord blood by assessment of the changes in brain from baseline in MRI on Day 7.
Intracranial Hemorrhage(MRI) | At the age of 12 months
  Efficacy of cord blood by assessment of the changes in brain from baseline in MRI on 12 months.
Number of Adverse Events | In 72 hours
  This is a composition of general appearance includes abdomen, skin, head and neck (including ears, eyes, nose, and throat), lymph nodes, thyroid, musculoskeletal and neurological systems.
Number of Adverse Events(Blood Pressure) | In 72 hours
  This is a composition of general appearance, blood pressure, pulse, respiratory, cardiovascular, abdomen, skin, head and neck (including ears, eyes, nose, and throat), lymph nodes, thyroid, musculoskeletal and neurological systems.
Number of Adverse Events(Pulse) | In 72 hours
  This is a composition of general appearance, blood pressure, pulse, respiratory, cardiovascular, abdomen, skin, head and neck (including ears, eyes, nose, and throat), lymph nodes, thyroid, musculoskeletal and neurological systems.
Number of Adverse Events(Respiratory) | In 72 hours
  This is a composition of general appearance, blood pressure, pulse, respiratory, cardiovascular, abdomen, skin, head and neck (including ears, eyes, nose, and throat), lymph nodes, thyroid, musculoskeletal and neurological systems.
Incidence of Complication | From birth to the age of 28 days in each treatment period
  To gain the incidence of Polycythemia, neutropenia, thrombocytopenia, hypertension, sepsis, intraventricular hemorrhage(IVH), periventricular leukomalacia(PVL), seizure, necrotizing enterocolitis (NEC), persistent ductus arterious (PDA), apnea of prematurity, pulmonary haemorrhage, pulmonary hypertension, Prolonged blood coagulation time, retinopathy of prematurity(ROP), cardiac arrhythmia, major venous thrombosis, Renal failure treated with dialysis, pneumonia, pulmonary airleak and chronic lung disease.
SDF-1 in Serum | At the age of 4 days
  Biomarkers for Oxidative Stress, Inflammation and immune response as a measure of efficacy for hypoxic ischemic encephalopathy or cerebral infarction.
SDF-1 in Serum | At the age of 14 days
  Biomarkers for Oxidative Stress, Inflammation and immune response as a measure of efficacy for hypoxic ischemic encephalopathy or cerebral infarction.
TNF-alpha in Serum | At the age of 4 days
  Biomarkers for Oxidative Stress, Inflammation and immune response as a measure of efficacy for hypoxic ischemic encephalopathy or cerebral infarction.
TNF-alpha in Serum | At the age of 14 days
  Biomarkers for Oxidative Stress, Inflammation and immune response as a measure of efficacy for hypoxic ischemic encephalopathy or cerebral infarction.
IL-1 in Serum | At the age of 4 days
  Biomarkers for Oxidative Stress, Inflammation and immune response as a measure of efficacy for hypoxic ischemic encephalopathy or cerebral infarction.
IL-1 in Serum | At the age of 14 days
  Biomarkers for Oxidative Stress, Inflammation and immune response as a measure of efficacy for hypoxic ischemic encephalopathy or cerebral infarction.

CONTACTS AND LOCATIONS:
Overall Officials: Wenhao Zhou, Doctor, Study Chair — Children's Hospital of Fudan University
Locations (1):
- Children Hospital of Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Cotten CM, Murtha AP, Goldberg RN, Grotegut CA, Smith PB, Goldstein RF, Fisher KA, Gustafson KE, Waters-Pick B, Swamy GK, Rattray B, Tan S, Kurtzberg J. Feasibility of autologous cord blood cells for infants with hypoxic-ischemic encephalopathy. J Pediatr. 2014 May;164(5):973-979.e1. doi: 10.1016/j.jpeds.2013.11.036. Epub 2013 Dec 31. PMID 24388332
- [Background] Walsh BH, Boylan GB, Livingstone V, Kenny LC, Dempsey EM, Murray DM. Cord blood proteins and multichannel-electroencephalography in hypoxic-ischemic encephalopathy. Pediatr Crit Care Med. 2013 Jul;14(6):621-30. doi: 10.1097/PCC.0b013e318291793f. PMID 23823198
- [Background] Walsh BH, Broadhurst DI, Mandal R, Wishart DS, Boylan GB, Kenny LC, Murray DM. The metabolomic profile of umbilical cord blood in neonatal hypoxic ischaemic encephalopathy. PLoS One. 2012;7(12):e50520. doi: 10.1371/journal.pone.0050520. Epub 2012 Dec 5. PMID 23227182
- [Background] Liao Y, Cotten M, Tan S, Kurtzberg J, Cairo MS. Rescuing the neonatal brain from hypoxic injury with autologous cord blood. Bone Marrow Transplant. 2013 Jul;48(7):890-900. doi: 10.1038/bmt.2012.169. Epub 2012 Sep 10. PMID 22964590
- [Background] Pimentel-Coelho PM, Rosado-de-Castro PH, da Fonseca LM, Mendez-Otero R. Umbilical cord blood mononuclear cell transplantation for neonatal hypoxic-ischemic encephalopathy. Pediatr Res. 2012 Apr;71(4 Pt 2):464-73. doi: 10.1038/pr.2011.59. Epub 2012 Feb 8. PMID 22430382
- [Background] Wiberg N, Kallen K, Herbst A, Olofsson P. Relation between umbilical cord blood pH, base deficit, lactate, 5-minute Apgar score and development of hypoxic ischemic encephalopathy. Acta Obstet Gynecol Scand. 2010 Oct;89(10):1263-9. doi: 10.3109/00016349.2010.513426. PMID 20846059